CLINICAL TRIAL: NCT03186313
Title: A Phase 3 Randomized, Open-Label, Study to Evaluate the Safety and Efficacy of the Combined Single Dose of Dactavira Plus (EPGCG, Sofosbuvir , Daclatasvir & Ribavirin) Versus Sofosbuvir + Daclatasvir + Ribavirin (Part A) and a Single Dose of Dactavira (EPGCG, Sofosbuvir & Daclatasvir) Versus Sofosbuvir + Daclatasvir (Part B) in Egyptian Adults With Chronic Genotype 4 HCV Infection
Brief Title: A Study to Evaluate the Safety and Efficacy of the Combined Single Dose of Dactavira Plus Or Dactavira in Egyptian Adults With Chronic Genotype 4 HCV Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Egyptian Liver Hospital (Other)
Collaborators: Wadi El Nil Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ELH - 2016
Record Dates: First submitted 2017-05-31; First posted 2017-06-14 (Actual); Last update posted 2017-12-27 (Actual); Status verified 2017-12

CONDITIONS: Hepatitis C
Keywords: HCV; Sofosbuvir; Ribavirin
MeSH Terms: conditions — Hepatitis C | interventions — Sofosbuvir; daclatasvir; Ribavirin

ARMS (4):
- Part A: Arm 1 (Experimental): Single daily dose (2 Tablets) of Dactavira Plus each tablet contains (EPGCG 200 mg , Sofosbuvir 200mg, Daclatasvir 30 mg, Ribavirin 400 mg) for 12 weeks.
  Interventions: Drug: Dactavira Plus
- Part A: Arm 2 (Active Comparator): Daily dose including Sofosbuvir 400 mg , Daclatasvir 60 mg & Ribavirin 800 mg for 12 weeks.
  Treatment assignments will be stratified according to the presence or absence of cirrhosis.
  Interventions: Drug: Sofosbuvir + Daclatasvir + Ribavirin
- Part B: Arm 3 (Experimental): Single daily dose (1 Tablet) of Dactavira each tablet contains (EPGCG 400 mg , Sofosbuvir 400mg, Daclatasvir 60 mg) for 12 weeks.
  Interventions: Drug: Dactavira
- Part B: Arm 4 (Active Comparator): Daily dose including Sofosbuvir 400 mg & Daclatasvir 60 mg for 12 weeks.
  Interventions: Drug: Sofosbuvir + Daclatasvir

INTERVENTIONS:
Drug: Dactavira Plus — 1 Single daily dose (2 Tablets) of Dactavira Plus each tablet contains (EPGCG 200 mg , Sofosbuvir 200mg, Daclatasvir 30 mg, Ribavirin 400 mg) for 12 weeks.
  Arms: Part A: Arm 1
Drug: Sofosbuvir + Daclatasvir + Ribavirin — Daily dose including Sofosbuvir 400 mg , Daclatasvir 60 mg & Ribavirin 800 mg for 12 weeks.
  Arms: Part A: Arm 2
Drug: Dactavira — Single daily dose (1 Tablet) of Dactavira each tablet contains (EPGCG 400 mg , Sofosbuvir 400mg, Daclatasvir 60 mg) for 12 weeks
  Arms: Part B: Arm 3
Drug: Sofosbuvir + Daclatasvir — Daily dose Sofosbuvir 400 mg & Daclatasvir 60 mg for 12 weeks
  Arms: Part B: Arm 4

SUMMARY:
A phase 3 Randomized, Open-Label, Study to Evaluate the Safety and Efficacy of the combined single dose of Dactavira Plus (EPGCG, Sofosbuvir , Daclatasvir & Ribavirin) versus Sofosbuvir + Daclatasvir + Ribavirin (Part A) and a single dose of Dactavira (EPGCG, Sofosbuvir & Daclatasvir) versus Sofosbuvir + Daclatasvir (Part B) in Egyptian Adults with Chronic Genotype 4 HCV Infection.

DETAILED DESCRIPTION:
Study Design: Part A Randomized, open-label study in treatment naïve cirrhotic adults with chronic genotype 4 HCV infection.

Treatment-naïve is defined as having never received treatment for HCV with any interferon (IFN), Ribavirin, or other approved or experimental HCV specific direct acting antivirals.

It is planned that 28 subjects will be enrolled in the study such that an approximate even number of treatment naïve subjects will be enrolled across the 2 treatment arms:

Arm 1 Single daily dose (2 Tablets) of Dactavira Plus each tablet contains (EPGCG 200 mg , Sofosbuvir 200mg, Daclatasvir 30 mg, Ribavirin 400 mg) for 12 weeks.

Arm 2 Daily dose including Sofosbuvir 400 mg , Daclatasvir 60 mg & Ribavirin 800 mg for 12 weeks.

Treatment assignments will be stratified according to the presence or absence of cirrhosis.

Diagnosis and Main Eligibility Criteria: HCV RNA > 104 IU/mL or HCV RNA > LLOQ and did not achieve SVR 12 after completing prior treatment in this study with chronic genotype 4 HCV infection. Treatment-naïve adults, male and non pregnant/non-lactating female subjects, ages 18 years or older.

Study Procedures/

Frequency: Study visits for all subjects will occur at screening, Baseline/Day 1. On-treatment visits will occur as follows:

* Part A, Arm 1 and 2 - at the end of Weeks 1, 2, 4, 8, 12.
* All subjects will complete a 4-Week Post-treatment visit regardless of treatment duration. Subjects with HCV RNA < LLOQ will continue to 12 Week Post treatment visits unless confirmed viral relapse occurs at which time subjects will be early terminated from the study.

Screening assessments include safety laboratory tests (chemistry, hematology, coagulation, and urinalysis), 12 lead ECG, HCV RNA, hemoglobin A1c, urine drug screen, liver imaging, serum B-hCG (for all female subjects of child-bearing potential), physical examination (with height and bodyweight), vital signs, medical history, concomitant medications, and adverse events.

On-treatment assessments include safety laboratory tests (chemistry, hematology, and coagulation), HCV RNA, urine pregnancy tests (for all female subjects of child-bearing potential), physical examination, vital signs, concomitant medications, and adverse events.

Post-treatment assessments include HCV RNA, urine pregnancy tests (for all female subjects of child-bearing potential), vital signs, concomitant medications, and adverse events.

Criteria for Evaluation:

Safety: Adverse events will be collected from baseline through the 4 Week Post-Treatment Visit and AEs related to study procedures, will be collected from when subjects sign the consent form. Clinical laboratory tests will be performed during treatment through the 12 Week Post-Treatment Visit.

Efficacy: Efficacy will be evaluated using scheduled assessments of HCV RNA performed using Gene Xpert HCV Test.

Statistical Methods: The primary efficacy endpoint is SVR12 (ie, HCV RNA < LLOQ 12 weeks post-treatment) in all subjects who are randomized and treated. No statistical hypothesis testing will be performed. For each of the two treatment groups, a 2-sided 95% confidence interval using the exact binomial distribution will be constructed.

All continuous endpoints will be summarized using an 8 number summary (n, mean, standard deviation, median, Q1, Q3, minimum, maximum) by treatment duration. All categorical endpoints will be summarized by number and percentage of subjects who meet the endpoint definition.

Safety endpoints will be analyzed by the number and percent of subjects with events or abnormalities for categorical values or using an 8 number summary (n, mean, standard deviation, median, Q1, Q3, minimum, maximum) for continuous data by treatment group.

This study will be conducted in accordance with the guidelines of Good Clinical Practices (GCPs) including archiving of essential documents.

Study Design: Part B

Randomized, open-label study in treatment naïve not cirrhotic adults with chronic genotype 4 HCV infection.

Treatment-naïve is defined as having never received treatment for HCV with any interferon (IFN), Ribavirin, or other approved or experimental HCV specific direct acting antivirals.

It is planned that 50 subjects will be enrolled in the study such that an approximate even number of treatment naïve subjects will be enrolled across the 2 treatment arms:

Arm 3 Single daily dose (1 Tablets) of Dactavira each tablet contains (EPGCG 400 mg , Sofosbuvir 400mg, Daclatasvir 60 mg) for 12 weeks.

Arm 4 Daily dose including Sofosbuvir 400 mg & Daclatasvir 60 mg for 12 weeks

Treatment assignments will be stratified according to the presence or absence of cirrhosis.

Diagnosis and Main Eligibility Criteria: HCV RNA > 104 IU/mL or HCV RNA > LLOQ and did not achieve SVR 12 after completing prior treatment in this study with chronic genotype 4 HCV infection. Treatment-naïve adults, male and non pregnant/non-lactating female subjects, ages 18 years or older.

Study Procedures/

Frequency: Study visits for all subjects will occur at screening, Baseline/Day 1. On-treatment visits will occur as follows:

At the end of Weeks 1, 2, 4, 8, 12.

All subjects will complete a 4-Week Post-treatment visit regardless of treatment duration. Subjects with HCV RNA < LLOQ will continue to 12 Week Post treatment visits unless confirmed viral relapse occurs at which time subjects will be early terminated from the study.

Screening assessments include safety laboratory tests (chemistry, hematology, coagulation, and urinalysis), 12 lead ECG, HCV RNA, hemoglobin A1c, urine drug screen, liver imaging, serum B-hCG (for all female subjects of child-bearing potential), physical examination (with height and bodyweight), vital signs, medical history, concomitant medications, and adverse events.

On-treatment assessments include safety laboratory tests (chemistry, hematology, and coagulation), HCV RNA, urine pregnancy tests (for all female subjects of child-bearing potential), physical examination, vital signs, concomitant medications, and adverse events.

Post-treatment assessments include HCV RNA, urine pregnancy tests (for all female subjects of child-bearing potential), vital signs, concomitant medications, and adverse events.

Criteria for Evaluation:

Safety: Adverse events will be collected from baseline through the 4 Week Post-Treatment Visit and AEs related to study procedures, will be collected from when subjects sign the consent form. Clinical laboratory tests will be performed during treatment through the 12 Week Post-Treatment Visit.

Efficacy: Efficacy will be evaluated using scheduled assessments of HCV RNA performed using Gene Xpert HCV Test.

Statistical Methods:

The primary efficacy endpoint is SVR12 (ie, HCV RNA < LLOQ 12 weeks post-treatment) in all subjects who are randomized and treated. No statistical hypothesis testing will be performed. For each of the two treatment groups, a 2-sided 95% confidence interval using the exact binomial distribution will be constructed.

All continuous endpoints will be summarized using an 8 number summary (n, mean, standard deviation, and median, Q1, Q3, minimum, maximum) by treatment duration. All categorical endpoints will be summarized by number and percentage of subjects who meet the endpoint definition.

Safety endpoints will be analyzed by the number and percent of subjects with events or abnormalities for categorical values or using an 8 number summary (n, mean, standard deviation, median, Q1, Q3, minimum, maximum) for continuous data by treatment group.

ELIGIBILITY:
Inclusion Criteria for Part A Subjects must meet the following inclusion criteria to be eligible for participation in this study.

1. Willing and able to provide written informed consent.
2. Male or female, age ≥ 18 years.
3. HCV RNA ≥ 104 IU/mL at screening.
4. Confirmed chronic HCV infection as documented by either:

   a. A positive anti-HCV antibody test or positive HCV RNA or positive HCV genotyping test at least 6 months prior to the Baseline/Day 1 visit.
5. HCV genotype 4 at screening as determined by the Central Laboratory. Any non definitive results will exclude the subject from study participation.

   a Presence of cirrhosis is defined as any one of the following:
   * Liver biopsy within 2 years of Screening showing cirrhosis
   * Fibroscan with a result of ≥ 12.5 kPa within 6 months of Baseline/Day1
6. Body mass index (BMI) ≥ 18 kg/m2.
7. Screening ECG without clinically significant abnormalities.
8. Subjects must have the following laboratory parameters at screening:

   * ALT ≤ 10 x the upper limit of normal (ULN)
   * AST ≤ 10 x ULN
   * Hemoglobin ≥ 12 g/dL for male, ≥ 11 g/dL for female subjects
   * Platelets > 50,000 cells/mm3
   * INR ≤ 1.5 x ULN unless subject has known hemophilia or is stable on an anticoagulant regimen affecting INR
   * Albumin ≥ 3 g/dL
   * Total Bilirubin ≤ 1.5 ULN
   * Creatinine clearance (CLcr) ≥ 60 mL/min, as calculated by the Cockcroft-Gault equation
9. Subject has not been treated with any investigational drug or device within 30 days of the screening visit.
10. A female subject is eligible to enter the study if it is confirmed that she is:

    a Not pregnant or nursing b Of non-childbearing potential (ie, women who have had a hysterectomy, both ovaries removed or medically documented ovarian failure, or are postmenopausal women > 50 years of age with cessation [for 12 months] of previously occurring menses), or c Of childbearing potential (ie, women who have not had a hysterectomy, both ovaries removed, or no medically documented ovarian failure). Women ≤ 50 years of age with amenorrhea will be considered to be of childbearing potential. These women must have a negative serum pregnancy test at screening and a negative urine pregnancy test on the Baseline/Day 1 visit prior to randomization. They must also agree to one of the following from 3 weeks prior to Baseline/Day 1 until 30 days after the last dose of treatment or 3 months after last dose of Ribavirin:

    • Complete abstinence from intercourse. Periodic abstinence from intercourse (eg, calendar, ovulation, symptothermal, post-ovulation methods) is not permitted.

    Or
    * Consistent and correct use of 1 of the following methods of birth control listed below in addition to a male partner who correctly uses a condom from the date of screening until 3 months after the last dose of Ribavirin. Women of childbearing potential must not rely on hormone-containing contraceptives as a form of birth control during the study. Female subjects using a hormone-containing contraceptive prior to screening may continue their contraceptive regimen in addition to the study specified methods of birth control.
    * Intrauterine device (IUD) with a failure rate of < 1% per year
    * Female barrier method: cervical cap or diaphragm with spermicidal agent
    * Tubal sterilization
    * Vasectomy in male partner
11. All male study participants must agree to consistently and correctly use a condom, while their female partner agrees to use either 1 of the non-hormonal methods of birth control listed above or a hormone-containing contraceptive listed below, from the date of screening until 7 months after their last dose of Ribavirin :

    • Implants of levonorgestrel
    * Injectable progesterone
    * Oral contraceptives (either combined or progesterone only)
    * Contraceptive vaginal ring
    * Transdermal contraceptive patch
12. Male subjects must agree to refrain from sperm donation for at least 6 months after the last dose of Ribavirin.
13. Subject must be of generally good health as determined by the Investigator.
14. Subject must be able to comply with the dosing instructions for study drug administration and able to complete the study schedule of assessments.

Inclusion Criteria for Part B Subjects must meet the following inclusion criteria to be eligible for participation in this study.

1. Willing and able to provide written informed consent.
2. Male or female, age ≥ 18 years.
3. HCV genotype 4 at screening as determined by the Central Laboratory. Any non definitive results will exclude the subject from study participation. Historical result from prior participation in this study is acceptable, if applicable.
4. Cohort 1 only: HCV RNA ≥ 104 IU/mL at screening.
5. Chronic HCV infection (≥ 6 months) documented by medical history.
6. HCV treatment naïve, defined as no prior exposure to any IFN, Ribavirin, or other approved or experimental HCV specific direct acting antiviral agent
7. BMI ≥ 18 kg/m2

   Absence of cirrhosis is defined as any one of the following:

   a Liver biopsy within 2 years of Screening showing absence of cirrhosis b Fibroscan with a result of ≤ 12.5 kPa within 6 months of Baseline/Day1 In the absence of a definitive diagnosis of the presence or absence of cirrhosis by the above criteria, a liver biopsy is required. Liver biopsy results supersede the results obtained by Fibroscan or FibroTest.
8. Screening ECG without clinically significant abnormalities.
9. Subjects must have the following laboratory parameters at screening:

   - ALT ≤ 10 x the upper limit of normal (ULN)

   - AST ≤ 10 x ULN

   - Hemoglobin ≥ 12 g/dL for male, ≥ 11 g/dL for female subjects

   - Platelets > 50,000 cells/mm3

   - INR ≤ 1.5 x ULN unless subject has known hemophilia or is stable on an anticoagulant regimen affecting INR
   * Albumin ≥ 3 g/dL
   * Total bilirubin ≤ 1.5 x ULN
   * Creatinine clearance (CLcr) ≥ 60 mL/min, as calculated by the Cockcroft-Gault equation Subjects who received prior treatment in this study and who currently do not fulfill all of the above requirements may be enrolled in Part B Cohort 2 at the request of the Investigator and with the approval of the Medical Monitor or Study Director.
10. Subject has not been treated with any investigational drug or device within 28 days of the Baseline/Day 1 visit.
11. A female subject is eligible to enter the study if it is confirmed that she is:

    d Not pregnant or nursing e Of non-childbearing potential (ie, women who have had a hysterectomy, both ovaries removed or medically documented ovarian failure, or are postmenopausal women > 50 years of age with cessation [for 12 months] of previously occurring menses), or f Of childbearing potential (ie, women who have not had a hysterectomy, both ovaries removed, or no medically documented ovarian failure). Women ≤ 50 years of age with amenorrhea will be considered to be of childbearing potential. These women must have a negative serum pregnancy test at screening and a negative urine pregnancy test on the Baseline/Day 1 visit prior to randomization. They must also agree to one of the following from 3 weeks prior to Baseline/Day 1 until 30 days after the last dose of treatment or 3 months after last dose of Ribavirin:

    • Complete abstinence from intercourse. Periodic abstinence from intercourse (eg, calendar, ovulation, symptothermal, post-ovulation methods) is not permitted.

    Or

    • Consistent and correct use of 1 of the following methods of birth control listed below in addition to a male partner who correctly uses a condom from the date of screening until 3 months after the last dose of Ribavirin. Women of childbearing potential must not rely on hormone-containing contraceptives as a form of birth control during the study. Female subjects using a hormone-containing contraceptive prior to screening may continue their contraceptive regimen in addition to the study specified methods of birth control.

    • Intrauterine device (IUD) with a failure rate of < 1% per year

    • Female barrier method: cervical cap or diaphragm with spermicidal agent

    • Tubal sterilization

    • Vasectomy in male partner
12. All male study participants must agree to consistently and correctly use a condom, while their female partner agrees to use either 1 of the non-hormonal methods of birth control listed above or a hormone-containing contraceptive listed below, from the date of screening until 7 months after their last dose of Ribavirin :

    * Implants of levonorgestrel
    * Injectable progesterone
    * Oral contraceptives (either combined or progesterone only)
    * Contraceptive vaginal ring
    * Transdermal contraceptive patch
13. Male subjects must agree to refrain from sperm donation for at least 6 months after the last dose of Ribavirin.
14. Subject must be of generally good health as determined by the Investigator.
15. Subject must be able to comply with the dosing instructions for study drug administration and able to complete the study schedule of assessments.

Exclusion Criteria:

1.2.1. Exclusion Criteria for Part A Subjects who meet any of the following exclusion criteria are not to be enrolled in this study.

1. Prior exposure to IFN, Ribavirin, or other approved or experimental direct-acting antiviral targeting the HCV.
2. Current or prior history of any of the following:

a Clinical hepatic decompensation (ie, ascites, encephalopathy or variceal hemorrhage) b Clinically-significant illness (other than HCV) or any other major medical disorder that may interfere with subject treatment, assessment or compliance with the protocol, or, current evaluation for a potentially clinically significant illness (other than HCV) c Gastrointestinal disorder or post operative condition that could interfere with the absorption of the study drug d Solid organ transplantation e Significant pulmonary disease, significant cardiac disease or porphyria f Psychiatric hospitalization, suicide attempt, and/or a period of disability as a result of their psychiatric illness within the last 5 years Subjects with psychiatric illness (without the prior mentioned conditions) that is well-controlled on a stable treatment regimen for at least 6 months prior to Baseline/Day 1 or that has not required medication in the last 12 months may be enrolled.

g Any malignancy within the 5 years prior to screening, with the exception of specific cancers that are cured by surgical resection (basal cell skin cancer, etc.), or current evaluation for possible malignancy h Difficulty with blood collection and/or poor venous access for the purposes of phlebotomy i 4. Infection with hepatitis B virus (HBV) or human immunodeficiency virus (HIV).

5. Contraindication to Ribavirin therapy e.g., history of clinically significant hemoglobinopathy (sickle cell disease, thalassemia).

6. History of malignancy diagnosed or treated within 5 years (recent localized treatment of squamous or non-invasive basal cell skin cancers is permitted; cervical carcinoma in situ is allowed if appropriately treated prior to screening); subjects under evaluation for malignancy are not eligible.

7. Chronic use of systemically administered immunosuppressive agents (eg, prednisone equivalent > 10 mg/day).

8. Clinically-relevant drug or alcohol abuse within 12 months of screening. A positive drug screen will exclude subjects unless it can be explained by a prescribed medication; the diagnosis and prescription should be approved by the investigator.

9. History of solid organ transplantation. 10. Current or prior history of clinical hepatic decompensation (eg, ascites, variceal hemorrhage, hepatic encephalopathy, hepatorenal syndrome and hepatopulmonary syndrome).

11. History of clinically-significant illness or any other major medical disorder that may interfere with subject treatment, assessment or compliance with the protocol.

12. History of a gastrointestinal disorder (or post-operative condition) that could interfere with the absorption of the study drug.

13. History of significant pulmonary disease, significant cardiac disease or porphyria.

14. Excessive alcohol ingestion, defined as 3 glasses/day (1 glass is equivalent to 284 mL beer, 125 mL wine, or 25 mL distilled spirits) for females and 4 glasses/day for males.

16. Known hypersensitivity to Ribavirin, the study investigational medicinal product, the metabolites, or formulation excipients.

1.2.2. Exclusion Criteria for Part B Subjects who meet any of the following exclusion criteria are not to be enrolled in this study.

1. Prior exposure to IFN, Ribavirin, or other approved or experimental direct-acting antiviral targeting the HCV.
2. Current or prior history of any of the following:

   a Clinically hepatic decompensation (ie, ascites, encephalopathy or variceal hemorrhage) b Clinically-significant illness (other than HCV) or any other major medical disorder that may interfere with subject treatment, assessment or compliance with the protocol, or, current evaluation for a potentially clinically significant illness (other than HCV) c Gastrointestinal disorder or post operative condition that could interfere with the absorption of the study drug d Solid organ transplantation e Significant pulmonary disease, significant cardiac disease or porphyria f Psychiatric hospitalization, suicide attempt, and/or a period of disability as a result of their psychiatric illness within the last 5 years Subjects with psychiatric illness (without the prior mentioned conditions) that is well-controlled on a stable treatment regimen for at least 6 months prior to Baseline/Day 1 or that has not required medication in the last 12 months may be enrolled.

   i Significant drug allergy (such as anaphylaxis or hepatotoxicity)
3. Chronic liver disease of a non-HCV etiology (eg, hemochromatosis, Wilson's disease, α1 antitrypsin deficiency, cholangitis)
4. Infection with hepatitis B virus (HBV) or human immunodeficiency virus (HIV)
5. Use of any prohibited concomitant medications
6. Contraindication to Ribavirin therapy, including significant history of clinically significant hemoglobinopathy (eg, sickle cell disease, thalassemia)
7. In the judgment of the investigatory, any clinically-relevant drug or alcohol abuse within 12 months of screening that may interfere with subject treatment, assessment of compliance with the protocol
8. Pregnant or nursing females or male with pregnant female partner
9. Known hypersensitivity to Sofosbuvir, or formulation excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
The primary efficacy endpoint is SVR12 (ie, HCV RNA < LLOQ 12 weeks post-treatment) | 12 weeks
  The primary efficacy endpoint is SVR12 (ie, HCV RNA < LLOQ 12 weeks post-treatment)

CONTACTS AND LOCATIONS:
Locations (1):
- Egyptian Liver Hospital, Sherbin, Dakahlia Governorate, Egypt

REFERENCES:
- [Background] Doss W, Shiha G, Hassany M, Soliman R, Fouad R, Khairy M, Samir W, Hammad R, Kersey K, Jiang D, Doehle B, Knox SJ, Massetto B, McHutchison JG, Esmat G. Sofosbuvir plus ribavirin for treating Egyptian patients with hepatitis C genotype 4. J Hepatol. 2015 Sep;63(3):581-5. doi: 10.1016/j.jhep.2015.04.023. Epub 2015 May 1. PMID 25937436
- See also: Egyptian Liver Hospital site — http://www2.mans.edu.eg/hosted/liver-ri/en/about_institute.htm